CLINICAL TRIAL: NCT01072539
Title: A Post-marketing Surveillance (Pms) Study Of Safety And Effectiveness In Patients With Tigecycline Treatment
Brief Title: Study Evaluating The Safety And Effectiveness In Subjects With Tigecycline Treatment
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: 3074X1-4527; B1811040 (Other: Alias Study Number)
Record Dates: First submitted 2010-02-17; First posted 2010-02-22 (Estimated); Results first posted 2016-05-30 (Estimated); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Complicated Skin and Skin Structure Infections; Complicated Intra-abdominal Infections; Community-Acquired Bacterial Pneumonia
Keywords: infection; Tygacil; PMS
MeSH Terms: conditions — Infections | interventions — Tigecycline

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients who have approved indications of Tygacil: Approved indications of Tygacil
  -complicated intraabdominal infection, complicated skin and skin structure infection, community-acquired bacterial pneumonia
  Interventions: Drug: tigecycline

INTERVENTIONS:
Drug: tigecycline — As prescribed by physician in usual clinical practice
  Other Names: Tygacil

SUMMARY:
The primary objective of this study is to identify any changes on the safety profile of adverse events and serious adverse events. And the secondary objective is to evaluate clinical response in the clinically evaluable population at test-of cure (TOC) or at the end of treatment (EOT) assessment, and microbiologic response at the subject level, if available.

DETAILED DESCRIPTION:
Prior to the conduct of this study, the investigator will explain the study objective, etc to prospective subjects on the basis of "explanatory material." The informed consent will be obtained in written form by each subject voluntarily.

ELIGIBILITY:
Inclusion Criteria:

Evidence of a personally signed and dated informed consent document indicating that the subject (or a legal representative) has been informed of all pertinent aspects of the study. Subjects must meet all of the following inclusion criteria to be eligible for enrollment into the study :

Adults 18 years of age or older, who have one of the followings:

* Complicated skin and skin structure infections
* Complicated intra-abdominal infections
* Community-acquired bacterial pneumonia

Exclusion Criteria:

Subjects presenting with any of the following will not be included in the study:

* Patients who have known hypersensitivity to tigecycline
* Patients with rare hereditary problems of galactose intolerance, the Lapp lactase deficiency, or glucose-galactose malabsorption

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: General Hospitals
Sampling Method: Non-Probability Sample
Enrollment: 3172 (Actual)
Dates: Start 2010-05; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (35):
- South Korea (35):
  - Ajou University Hospital, Suwon, Gyeonggi-do
  - Pusan National University Yangsan Hospital, Yangsan, Gyeongsangnam-do
  - Gachon University Gil Hospital, Namdong-gu, Incheon
  - Wonkwang University Hospital, Iksan-si, Jeollabuk-do
  - Chonbuk National University Hospital, Jeonju, Jeollabuk-do
  - Hanil Medical Center, Dobong-Gu, Seoul
  - Kosin University Gospel Hospital, Busan
  - Dong-A University Medical Center (Dong-A University Hospital), Busan
  - Cheongju St. Mary's Hospital, Cheongju-si
  - Keimyung University Dongsan Medical Center (KUDMC), Daegu
  - Kyungpook National University Hospital (KNUH), Daegu
  - Daegu fatima hospital, Daegu
  - Yeungnam University Medical Center, Daegu
  - Daegu Catholic University Medical Center (DCUMC), Daegu
  - Korea University Ansan Hospital, Gyeonggi-do
  - Ajou University Hospital, Gyeonggi-do
  - Inha University Hospital, Incheon
  - Gachon University Gil Hospital, Incheon
  - Jeju National University Hospital, Jeju City
  - Yonsei University Wonju College of Medicine- Wonju Christian Hospital, Kangwon-do
  - Korea University Anam Hospital, Seoul
  - Yonsei University College of Medicine Severance Hospital Rheumatology Internal Medicine, Seoul
  - Kyunghee University Medical Hospital, Seoul
  - Hallym University Kangdong Sacred Heart Hospital, Seoul
  - Kyung Hee University Hospital at Gangdong, Seoul
  - Kangdong Sacred Heart Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Asan Medical Center, University of Ulsan, Seoul
  - Asan Medical Center, Seoul
  - Eulji Medical Center, Seoul
  - Hallym University Kangnam Sacred Heart Hospital, Seoul
  - Hallym University Medical Center (HUMC) - Kangnam Sacred Heart Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Kangbuk Samsung Medical Center, Seoul
  - Ulsan University Hospital, Ulsan

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=3074X1-4527&StudyName=Study%20Evaluating%20The%20Safety%20And%20Effectiveness%20In%20Subjects%20With%20Tigecycline%20Treatment

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled between May 2010 and April 2015 from Korean health care centers.
Groups:
- Tygacil: Participants were administered Tygacil as part of routine practice. The use and dosage recommendations for Tygacil were based on the approved local product document and were adjusted solely according to medical and therapeutic necessity.
Period: Overall Study
Arm/Group | Tygacil
Started | 3172
Completed | 3169 (Refer to the Safety Analysis Set. Data for completion were not collected.)
Not Completed | 3
Not completed — Treated prior to the Site Initiation | 1
Not completed — Protocol Violation | 2

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: participants who received at least one dose of Tygacil and had related safety endpoints evaluated at least once.
Arm/Group | Tygacil
Number analyzed (Participants) | 3169
Age, Customized [Number; unit: Participants]
  <30 years | 126
  30 to 39 years | 200
  40 to 49 years | 346
  50 to 64 years | 1116
  >=65 years | 1381
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1089
  Male | 2080
Infection Site [Number; unit: Participants] — cSSSI: Complicated skin and skin structure infection; cIAI: Complicated intra-abdominal infection; CAP: Community-acquired bacterial pneumonia.
  Participants
    cSSSI | 976
    cIAI | 1947
    CAP | 242
    cIAI + cSSSI | 2
    cIAI + CAP | 2
Severity of Infection [Number; unit: Participants]
  Mild | 287
  Moderate | 2072
  Severe | 810

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Adverse Events (AEs)/Adverse Drug Reactions (ADRs), Serious AEs (SAEs)/Serious ADRs (SADRs), and Unexpected AEs/ADRs
Description: All AEs reported after start of administration of Tygacil were considered as on treatment and summarized. All AEs, except for those with causal relationship to the study drug assessed as "unlikely", were considered as ADRs. Unexpected AEs/ADRs were classified by medical review with reference to the approved local product document and confirmed by Pfizer.
Time Frame: From the time of the participant's first dosing in the observational period as per study design through and including 28 calendar days after the last administration of the study drug within the observational period.
Population: Safety Analysis Set
Measure: Number; unit: Percentage of Participants
Arm/Group | Tygacil
Number analyzed (Participants) | 3169
Percentage of Participants
  AEs | 32.98
  ADRs | 9.85
  SAEs | 13.22
  SADRs | 0.13
  Unexpected AEs | 8.24
  Unexpected ADRs | 0.44

2. Secondary Outcome: Percentage of Participants With Clinical Response of Cure or Improvement at the Test-of-Cure(TOC) or End-of-Treatment (EOT) Assessment
Description: Participants whose clinical response was assessed as cure or improvement at the TOC or EOT assessment were considered as "effective" to the treatment of Tygacil .
Time Frame: At the TOC or EOT assessment
Population: Effectiveness Analysis Set: Participants who received at least one dose of Tygacil and had related effectiveness endpoints evaluated at least.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Tygacil
Number analyzed (Participants) | 2545
Percentage of Participants
  Prospectively Collected Data | 59.68 [55.63 to 63.73]
  Retrospectively Collected Data | 74.97 [73.07 to 76.88]
  Total | 71.59 [69.84 to 73.34]

3. Secondary Outcome: Percentage of Participants With Clinical Response of Cure or Improvement at the TOC or EOT Assessment by Infection Site
Description: as for outcome 2
Time Frame: At the TOC or EOT assessment
Population: Effectiveness Analysis Set.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Tygacil
Number analyzed (Participants) | 2545
Percentage of Participants
  Infection Site: cSSSI | 77.53 [74.66 to 80.41]
  Infection Site: cIAI | 71.52 [69.28 to 73.76]
  Infection Site: CAP | 45.35 [37.91 to 52.79]
  Infection Site: cIAI + cSSSI | 0.00 [0.00 to 0.00]
  Infection Site: cIAI + CAP | 50.00 [0.00 to 100.00]
  Infection Site: Total | 71.59 [69.84 to 73.34]
Statistical Analysis 1: Comparison: Tygacil; Comparison among subgroups of Infection Sites: cSSSI, cIAI, CAP, cIAI + cSSSI, and cIAI + CAP; Test type: Superiority or Other; p < 0.0001, Fisher Exact — Statistical significant level: 0.05

4. Primary Outcome: Percentage of Participants With Adverse Events by Baseline and Treatment Characteristics
Description: Baseline and treatment characteristics included: prospectively/retrospectively collected data, geriatric status (<65 years or >=65 years), age categories, sex, duration of disease, infection site, severity of infection, general, present and past medical history, kidney disorder, liver disorder, total administration period of Tygacil, mean daily dose of Tygacil, past medication and therapy, and concomitant medications.
Time Frame: as for outcome 1
Population: Safety Analysis Set.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Tygacil
Number analyzed (Participants) | 3169
Percentage of Participants
  Prospectively Collected Data | 34.15 [30.73 to 37.57]
  Retrospectively Collected Data | 32.62 [30.76 to 34.48]
  Geriatric: <65 Years | 30.98 [28.84 to 33.13]
  Geriatric: >=65 Years | 35.55 [33.03 to 38.08]
  Age: <30 Years | 30.16 [22.15 to 38.17]
  Age: 40 to 49 Yeas | 27.46 [22.75 to 32.16]
  Age: 50 to 64 Years | 31.99 [29.25 to 34.73]
  Age: >=65 Years | 35.55 [33.03 to 38.08]
  Sex: Male | 32.55 [30.53 to 34.56]
  Sex: Female | 33.79 [30.98 to 36.60]
  Duration of Disease: <3 Months | 32.88 [31.15 to 34.60]
  Duration of Disease: >=3 Months and <6 Months | 33.63 [27.43 to 39.83]
  Duration of Disease: >=6 Months | 32.20 [20.28 to 44.13]
  Infection Site: cSSSI | 28.79 [25.95 to 31.63]
  Infection Site: cIAI | 34.87 [32.76 to 36.99]
  Infection Site: CAP | 34.30 [28.32 to 40.28]
  Infection Site: cIAI + cSSSI | 50.00 [0.00 to 100.00]
  Infection Site: cIAI + CAP | 50.00 [0.00 to 100.00]
  Severity of Infection: Mild | 26.83 [21.70 to 31.96]
  Severity of Infection: Moderate | 27.27 [25.35 to 29.19]
  Severity of Infection: Severe | 49.75 [46.31 to 53.20]
  General Medical History: Yes | 34.91 [33.19 to 36.63]
  General Medical History: No | 6.48 [3.20 to 9.76]
  General Medical History (Present): Yes | 35.03 [33.29 to 36.76]
  General Medical History (Present): No | 9.45 [5.85 to 13.05]
  General Medical History (Past): Yes | 37.10 [34.14 to 40.05]
  General Medical History (Past): No | 31.00 [29.04 to 32.96]
  Kidney Disorder: Yes | 46.86 [42.89 to 50.84]
  Kidney Disorder: No | 29.69 [27.92 to 31.46]
  Liver Disorder: Yes | 39.82 [36.65 to 43.00]
  Liver Disorder: No | 30.20 [28.30 to 32.09]
  Total Treatment Period of Tygacil: <7 Days | 34.74 [31.40 to 38.09]
  Total Treatment Period of Tygacil: 7 to 14 Days | 29.94 [27.39 to 32.49]
  Total Treatment Period of Tygacil: >14 Days | 34.99 [32.23 to 37.74]
  Mean Daily Dose of Tygacil: <50 mg | 100.00 [100.00 to 100.00]
  Mean Daily Dose of Tygacil: 50 to <100 mg | 39.92 [36.50 to 43.35]
  Mean Daily Dose of Tygacil: 100 to <200 mg | 30.57 [28.72 to 32.42]
  Mean Daily Dose of Tygacil: >=200 mg | 60.00 [17.06 to 100.00]
  Past Medication and Therapy: Yes | 33.48 [31.77 to 35.19]
  Past Medication and Therapy: No | 27.02 [21.49 to 32.54]
  Concomitant Medications: Yes | 33.77 [32.09 to 35.45]
  Concomitant Medications: No | 14.06 [8.04 to 20.08]
Statistical Analysis 1: Comparison: Tygacil; Geriatrc: <65 Years Versus (VS) Geriatrc: >=65 Years; Test type: Superiority or Other; p = 0.0067, Chi-squared — Statistical significant level: 0.05
Statistical Analysis 2: Comparison: Tygacil; Comparison among Age categories: <30 Years, 30 to 39 Years, 40 to 49 Years, 50 to 64 Years, and >=65 Years; Test type: Superiority or Other; p = 0.0412, Chi-squared — Statistical significant level: 0.05
Statistical Analysis 3: Comparison: Tygacil; Sex: Male VS Sex: Female; Test type: Superiority or Other; p = 0.4792, Chi-squared — Statistical significant level: 0.05
Statistical Analysis 4: Comparison: Tygacil; Comparson among Duration of Disease categories: <3 Months, >=3 Months and <6 Months, and >=6 Months; Test type: Superiority or Other; p = 0.9669, Chi-squared — Statistical significant level: 0.05
Statistical Analysis 5: Comparison: Tygacil; Comparison among subgroups of infection site: cSSSI, cIAI, CAP, cIAI + cSSSI, and cIAI + CAP; Test type: Superiority or Other; p = 0.0064, Fisher Exact — Statistical significant level: 0.05
Statistical Analysis 6: Comparison: Tygacil; Comparison among severity of infection subgroups: Mild, Moderate, and Severe; Test type: Superiority or Other; p < 0.0001, Chi-squared — Satistical significant level: 0.05
Statistical Analysis 7: Comparison: Tygacil; General Medical History: Yes VS General Medical History: No; Test type: Superiority or Other; p < 0.0001, Chi-squared — Statistical significant level: 0.05
Statistical Analysis 8: Comparison: Tygacil; General Medical History (Present): Yes VS General Medical History (Present): No; Test type: Superiority or Other; p < 0.0001, Chi-squared — Statistical significant level: 0.05
Statistical Analysis 9: Comparison: Tygacil; General Medical History (Past): Yes VS General Medical History (Past): No; Test type: Superiority or Other; p = 0.0006, Chi-squared — Statistical significant level: 0.05
Statistical Analysis 10: Comparison: Tygacil; Kidney Disorder: Yes VS Kidney Disorder: No; Test type: Superiority or Other; p < 0.0001, Chi-squared
Statistical Analysis 11: Comparison: Tygacil; Liver Disorder: Yes VS Liver Disorder: No; Test type: Superiority or Other; p < 0.0001, Chi-squared — Statistical significant level: 0.05
Statistical Analysis 12: Comparison: Tygacil; Comparison among subgroups of Total Treatment Period of Tygacil: <7 Days, 7 to 14 Days, and >14 Days; Test type: Superiority or Other; p = 0.0153, Chi-squared — Statistical significant level: 0.05
Statistical Analysis 13: Comparison: Tygacil; Comparison among subgroups of Mean Daily Dose of Tygacil: <50 mg, 50 to <100 mg, 100 to <200 mg, and >=200 mg; Test type: Superiority or Other; p < 0.0001, Fisher Exact — Statistical significant level 0.05
Statistical Analysis 14: Comparison: Tygacil; Past Medication and Therapy: Yes VS Past Medication and Therapy: No; Test type: Superiority or Other; p = 0.0376, Chi-squared — Statistical significant level: 0.05
Statistical Analysis 15: Comparison: Tygacil; Concomitant Medications: Yes VS Concomitant Medications: No; Test type: Superiority or Other; p < 0.0001, Chi-squared — Statistical significant level: 0.05

5. Secondary Outcome: Percentage of Participants by Microbiologic Response at the Participant Level (Prospective Study Phase)
Description: Definitions: Eradication: None of the baseline isolates were present in a repeat culture taken from the original site of infection (documented) or a clinical response of cure precluded the availability of a specimen for culture (presumed). Persistence: Any baseline isolates were present in a repeat culture obtained from the original site of infection (documented) or culture data were not available for a participant with a clinical response of failure (presumed). Unevaluable: participants who died during therapy for non-infection-related reasons, died for any reason within 2 days after first administration of Tygacil, were lost to follow-up (ie, clinical response was not able to be assessed), or had no baseline isolates.
Time Frame: At the TOC or EOT assessment
Population: Effectiveness Analysis Set from the prospective study phase; n refers to the total nunber of participants who had evaluable data.
Measure: Number; unit: Percentage of Participants
Arm/Group | Tygacil
Number analyzed (Participants) | 563
Percentage of Participants
  Eradication (Documented or Presumed) (n=514) | 46.69
  Persistence (Documented or Presumed) (n=514) | 32.68
  Unevaluable (n=514) | 20.62

ADVERSE EVENTS:
Time Frame: From the time of the participant's first dosing in the observational period as per study design through and including 28 calendar days after the last administration of the study drug within the observational period.
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Tygacil
Serious Adverse Events (participants affected / at risk) | 419/3169
Other Adverse Events (participants affected / at risk) | 537/3169
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tygacil (N=3169)
Exacerbation of disease (General disorders) | 1
Mediastinitis (General disorders) | 2
Multiple organ failure (General disorders) | 33
Cardiac failure (Cardiac disorders) | 5
Circulatory failure (Vascular disorders) | 3
Hypotension (Vascular disorders) | 7
Brain hypoxia (Nervous system disorders) | 2
Brain stem disorder (Nervous system disorders) | 1
Carboxyhaemoglobinaemia (Nervous system disorders) | 1
Convulsions (Nervous system disorders) | 2
Oedema cerebral (Nervous system disorders) | 1
Clostridial infection (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Colitis pseudomembranous (Gastrointestinal disorders) | 1
Gastric ulcer haemorrhagic (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2
Intestinal fistula (Gastrointestinal disorders) | 1
Intestinal ischaemia (Gastrointestinal disorders) | 1
Intestinal perforation (Gastrointestinal disorders) | 1
Melaena (Gastrointestinal disorders) | 2
Pancreatitis (Gastrointestinal disorders) | 3
Arrhythmia (Cardiac disorders) | 2
Bradycardia (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 4
Fibrillation atrial (Cardiac disorders) | 3
Fibrillation ventricular (Cardiac disorders) | 1
Sick sinus syndrome (Cardiac disorders) | 1
Bilirubinaemia (Hepatobiliary disorders) | 2
Cholangitis (Hepatobiliary disorders) | 3
Cholelithiasis (Hepatobiliary disorders) | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 5
Hepatic failure (Hepatobiliary disorders) | 11
Hepatic function abnormal (Hepatobiliary disorders) | 1
Hepatitis (Hepatobiliary disorders) | 1
Hepatocellular damage (Hepatobiliary disorders) | 1
Hepatorenal syndrome (Hepatobiliary disorders) | 3
Jaundice (Hepatobiliary disorders) | 2
Serum glutamic oxaloacetic transaminase increased (Hepatobiliary disorders) | 3
Serum glutamic pyruvate transaminase increased (Hepatobiliary disorders) | 2
Acidosis (Metabolism and nutrition disorders) | 1
Myositis (Musculoskeletal and connective tissue disorders) | 1
Cardiomyopathy (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 4
Myocardial ischaemia (Cardiac disorders) | 1
Carcinoma small intestine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Leukaemia granulocytic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Melanoma malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 45
Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Coagulation disorder (Blood and lymphatic system disorders) | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 5
Haemorrhage not otherwise specified (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 8
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Chronic obstructive airways disease (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 47
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 3
Respiratory insufficiency (Respiratory, thoracic and mediastinal disorders) | 7
Respiratory tract haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Diabetic ulcer (Skin and subcutaneous tissue disorders) | 1
Stevens johnson syndrome (Skin and subcutaneous tissue disorders) | 2
Azotaemia (Renal and urinary disorders) | 3
Renal failure acute (Renal and urinary disorders) | 10
Renal failure chronic (Renal and urinary disorders) | 1
Renal failure chronic aggravated (Renal and urinary disorders) | 8
Renal function abnormal (Renal and urinary disorders) | 3
Cerebral haemorrhage (Vascular disorders) | 1
Cerebral infarction (Vascular disorders) | 1
Haematoma (Vascular disorders) | 2
Thrombophlebitis deep (Vascular disorders) | 1
Leucopenia (Blood and lymphatic system disorders) | 1
Leukocytosis (Blood and lymphatic system disorders) | 1
Marrow depression (Blood and lymphatic system disorders) | 6
Pancytopenia (Blood and lymphatic system disorders) | 1
Graft versus host disease (Immune system disorders) | 1
Application site reaction (Injury, poisoning and procedural complications) | 1
Cellulitis (Infections and infestations) | 1
Abscess (Infections and infestations) | 8
Infection aggravated (Infections and infestations) | 3
Peritonitis (Infections and infestations) | 6
Pyelonephritis (Renal and urinary disorders) | 1
Sepsis (Infections and infestations) | 139
Wound dehiscence (Injury, poisoning and procedural complications) | 1
Amputation (Surgical and medical procedures) | 2
Secondary carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Surgical intervention (Surgical and medical procedures) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tygacil (N=3169)
Diarrhoea (Gastrointestinal disorders) | 45
Nausea (Gastrointestinal disorders) | 170
Vomiting (Gastrointestinal disorders) | 42
Serum glutamic oxaloacetic transaminase increased (Hepatobiliary disorders) | 72
Serum glutamic pyruvate transaminase increased (Hepatobiliary disorders) | 62
Phosphatase alkaline increased (Metabolism and nutrition disorders) | 42
Thrombocytopenia (Blood and lymphatic system disorders) | 38
Azotaemia (Renal and urinary disorders) | 66

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.